CLINICAL TRIAL: NCT03240536
Title: Choosing Tests Wisely in Rheumatology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 109363
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: SLE
Keywords: Rheumatology Referral; Choosing Wisely

STUDY DESIGN:
Intervention Model Description: Randomized Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Ordering physicians who have referred to a rheumatologist in the St. Joseph's rheumatology clinic randomized to the intervention group will receive a brief Choosing Wisely form (for education of guidelines) faxed with the referral notice. At one and two years all ordering physicians will receive by fax a three question survey.
  Interventions: Other: Choosing Wisely form
- Control Group (No Intervention): Ordering physicians who have referred to rheumatologists in the control group will not receive the Choosing Wisely form. At one and two years all ordering physicians will receive by fax a three question survey.

INTERVENTIONS:
Other: Choosing Wisely form — The investigators will fax a "Choosing Wisely form" to ordering physicians that will include information from the Canadian Rheumatology Association Canada Choosing Wisely Guidelines. Three points will be included with some additional explanation of why these are important.
  The three guidelines included will be:
  1. Don't order an ANA as a screening test in patients without specific signs or symptoms of systemic lupus erythematous (SLE) or another connective tissue disorder (CTD).
  2. Don't routinely image patients with low back pain regardless of the duration of symptoms unless that are clinical reasons to suspect serious underlying pathology
  3. Don' routinely order a shoulder ultrasound as it is likely to indicate a tear in many people over the age of 50 years and will not change the initial management.
  Arms: Intervention Group

SUMMARY:
This is a randomized study intended to produce a reduction in ordering of inappropriate tests by general practitioners as determined by recommendations from the CRA's Choosing Wisely guidelines. This reduction of inappropriate testing is expected in referrals to the rheumatologists randomized to the intervention group. This study will further explore which recommendations from the Canadian Rheumatology Association (CRA)/Canada Choosing Wisely campaign have the most impact on regional referring physicians to the Rheumatology clinic at St. Joseph's Hospital, London.

DETAILED DESCRIPTION:
This a randomized study in that 6 rheumatologists (30 referrals each) will be randomized to one of two groups: intervention or control. Referring physicians to the intervention group will be faxed a brief Choosing Wisely form (intervention) based upon the recommendations of the Canadian Rheumatology Association's (CRA) Canada Choosing Wisely campaign, while referring physicians from the control group will not receive the form (non intervention). Analysis will be based upon the results of a three question survey faxed to all referring physicians at year one and at year two and on future referrals from the referring physicians to determine if there is a reduction in the group of ordering physicians that received the intervention (Choosing Wisely form).

ELIGIBILITY:
Inclusion Criteria:

* Ordering physicians who recently made a referral to the Rheumatology clinic at St. Joseph's Health Care.

Exclusion Criteria:

* N/A, all recent referrals will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Assessing the change in the number of the total number of ANA tests, back CT's and shoulder ultrasounds in rheumatology referrals | Change from baseline number of tests at year one, year two
  -collecting the total number of ANA tests, back CT's and shoulder ultrasounds

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No